CLINICAL TRIAL: NCT03516942
Title: Longitudinal Assessment of Financial Burden in Patients With Colon or Rectal Cancer Treated With Curative Intent
Brief Title: Financial Burden Assessment in Patients With Stage I-III Colon or Rectal Cancer Undergoing Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: EAQ162CD; NCI-2018-00151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ162CD (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAQ162CD (Other: DCP); ECOG-ACRIN-EAQ162CD (Other: CTEP); U10CA180820 (NIH); UG1CA189828 (NIH)
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Stage I Colon Cancer AJCC v8; Stage I Rectal Cancer AJCC v8; Stage II Colon Cancer AJCC v8; Stage II Rectal Cancer AJCC v8; Stage IIA Colon Cancer AJCC v8; Stage IIA Rectal Cancer AJCC v8; Stage IIB Colon Cancer AJCC v8; Stage IIB Rectal Cancer AJCC v8; Stage IIC Colon Cancer AJCC v8; Stage IIC Rectal Cancer AJCC v8; Stage III Colon Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Colon Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients complete questionnaires over 20-60 minutes at baseline and at 3, 6, 12, and 24 months after cancer diagnosis.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies the financial burden in patients with stage I-III colon or rectal cancer who are undergoing treatment. Collecting data from patients about their cost and quality of life may help doctors to better understand the impact of cancer treatment on a patient?s employment and finances.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the change in level of self-reported financial burden from baseline (within 60 days of diagnosis) to 12 months after diagnosis of colon or rectal cancer treated with curative-intent.

SECONDARY OBJECTVIES:

I. Evaluate reported access and utilization of financial services (i.e. financial counselor, navigator, social workers) and its association to financial burden in the first 12 months after diagnosis of colon or rectal cancer treated with curative-intent.

II. Evaluate the change in level of self-reported financial burden and employment limitations from baseline (within 60 days of diagnosis) to 3, 6, and 12 months after diagnosis of colon or rectal cancer treated with curative-intent.

III. Evaluate long term outcomes at 24 months after diagnosis including financial burden, employment limitations and adherence to clinical follow-up guidelines.

IV. Evaluate the change of quality-of-life outcome (QoL) from baseline to 12 months and its association with predictors.

V. Evaluate the change in level of self-reported financial burden from baseline to 12 months using alternate measures of financial burden (i.e. impact of cost questions and single item from European Organization for Research and Treatment of Cancer [EORTC] questionnaire [Q]30).

OUTLINE:

Patients complete questionnaires over 20-60 minutes at baseline and at 3, 6, 12, and 24 months after cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a life expectancy of >= 24 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3
* Patients must have a newly diagnosed colon or rectal cancer (initial diagnosis, either a biopsy or curative surgery, whichever is most recent) within 60 days of registration and have not yet received radiation or chemotherapy
* Patients must have stage I, II, or III disease at the time of enrollment and will be treated with curative-intent; this can be defined either clinically or pathologically if they have already undergone surgery; for staging of both colon and rectal cancer, the definition of stage I-III is based on the seventh edition (2010) or an updated version of the tumor, node, metastasis (TNM) staging system
* Patients are not eligible if they are already enrolled on a treatment clinical trial at the time of registration; they can remain on the study if they subsequently enroll on a treatment clinical trial during the study time period
* Patients who choose to not receive radiation and/or chemotherapy after a curative-intent surgery are eligible to participate
* Patients with a history of previous malignancy (except non-melanoma skin or cervical in-situ cancer) treated (with either surgery, chemotherapy, and/or radiation) within the last 3 years are not eligible
* Patients must be able to complete questionnaires in English
* Patients must sign and give written informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from a gastroenterology, surgical oncology, radiation oncology, or medical oncology clinic with newly diagnosed colon or rectal cancer are potential candidates for the study. Subjects must enroll within 60 days of their diagnostic biopsy or curative-intent surgery and prior to any chemotherapy and/or radiation
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2028-09-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sheetal Kircher, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (716):
- United States (716):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - CarolinaEast Oncology and Hematology Associates, New Bern, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Oncology Specialists-Statesville, Stateville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Sadigh G, Duan F, An N, Gareen ID, Sicks J, Suga JM, Kehn H, Mehan PT, Bajaj R, Hanson DS, Dalia SM, Acoba JD, Yasar DG, Taylor MA, Park E, Wagner LI, Kircher SM, Carlos RC. Financial Hardship Among Patients With Early-Stage Colorectal Cancer. JAMA Netw Open. 2024 Sep 3;7(9):e2431967. doi: 10.1001/jamanetworkopen.2024.31967. PMID 39287948
- [Derived] Kircher S, Duan F, An N, Gareen IF, Sicks JD, Sadigh G, Suga JM, Kehn H, Mehan PT, Bajaj R, Hanson DS, Dalia SM, Acoba JD, Yasar DG, Park ER, Wagner LI, Carlos RC. Patient-Reported Financial Burden of Treatment for Colon or Rectal Cancer. JAMA Netw Open. 2024 Jan 2;7(1):e2350844. doi: 10.1001/jamanetworkopen.2023.50844. PMID 38194233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a, longitudinal cohort study of financial burden in patients with colon, rectal, or rectosigmoid junction cancer. Measurements of financial burden (COST score) were collected at 5 time points over a 24-month follow-up period. Surveys were completed both by sites, to identify available clinical resources, and by participants, to assess the QoL and cost.
  The primary endpoint of this study was the change of the COST score from the baseline measurement to the 12-month follow-up (FU).
Groups:
- Observational (Questionnaire): Patients submitted questionnaires assessing financial burden
Period: Registration through baseline survey com
Arm/Group | Observational (Questionnaire)
Started | 565
Activated Surveys | 463
Completed | 463
Not Completed | 102
Not completed — Withdrawal by Subject | 36
Not completed — Death | 8
Not completed — Could not contact patient after enrollment | 58
Period: T0: Baseline
Arm/Group | Observational (Questionnaire)
Started | 463
Submitted T0 baseline survey | 450
Completed | 450
Not Completed | 13
Not completed — LOST | 13
Period: T1: 3 Months Survey
Arm/Group | Observational (Questionnaire)
Started | 450 (All participants completing the baseline survey have the opportunity to complete a survey at each timepoint. That is, failure to complete a survey (other than the baseline) in a prior period does not preclude completion of the survey in the current period.)
Submitted T0 and T1 surveys | 264
Completed | 264
Not Completed | 186
Not completed — Withdrawal by Subject | 13
Not completed — Death | 10
Not completed — Lost | 163
Period: T2: 6 Month Survey
Arm/Group | Observational (Questionnaire)
Started | 450 (All participants completing the baseline survey have the opportunity to complete a survey at each timepoint. That is, failure to complete a survey (other than the baseline) in a prior period does not preclude completion of the survey in the current period.)
Completed T0 and T2 surveys | 241
Completed T0, T1, and T2 surveys | 203
Completed | 241
Not Completed | 209
Not completed — Withdrawal by Subject | 15
Not completed — Death | 14
Not completed — Lost | 180
Period: T3: 12 Month Survey
Arm/Group | Observational (Questionnaire)
Started | 450 (All participants completing the baseline survey have the opportunity to complete a survey at each timepoint. That is, failure to complete a survey (other than the baseline) in a prior period does not preclude completion of the survey in the current period.)
Completed T0 and T3 surveys | 207
Completed T0, T1, T2 and T3 surveys | 151
Completed | 207
Not Completed | 243
Not completed — Withdrawal by Subject | 15
Not completed — Death | 19
Not completed — Lost | 209

BASELINE CHARACTERISTICS:
Population: Baseline characteristics reported for individual completing the baseline survey
Groups:
- Observational (Questionnaire): Patients complete questionnaires to assess financial burden
Arm/Group | Observational (Questionnaire)
Number analyzed (Participants) | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210
  Male | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 424
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 33
  White | 379
  More than one race | 4
  Unknown or Not Reported | 5
Employment [Count of Participants; unit: Participants]
  Employed | 214
  Retired | 153
  Unemployed | 77
  Not Answered | 6
Cancer Type [Count of Participants; unit: Participants]
  Colon Cancer | 289
  Rectal Cancer | 140
  Rectosigmoid Junction | 21
Cancer Stage at Enrollment [Count of Participants; unit: Participants] — This can be defined either clinically or pathologically if they have already undergone surgery. For staging of both colon and rectal cancer, the definition of stage I-III is based on the seventh edition (2010) or an updated version of the TNM staging system.
  Higher stage indicates more advanced disease as defined int he TNM staging system.
  Participants
    Stage l | 68
    Stage lI | 140
    Stage III | 242
Chemotherapy [Count of Participants; unit: Participants]
  Schedule Chemotherapy | 267
  No Chemtherapy | 183

OUTCOME MEASURES:

1. Primary Outcome: Comprehensive Score for Financial Toxicity (COST)
Description: The Comprehensive Score for Financial Toxicity (COST) COST is an 11-item patient-reported outcome (PRO) of financial hardship that uses a 7-day time window and 5-point Likert response scale (ranging from 0, indicating not at all, to 4, very much). Higher COST scores (range, 0-44) represent better financial well-being.
  The primary objective is to evaluate the change in the level of self-reported financial burden from baseline (within 60 days of diagnosis) to 12 months from study registration. (12 mo - baseline)
Time Frame: Baseline and 12 months after cancer diagnosis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- T0: Observational (Questionnaire): Patients with complete questionnaires to assess financial burden at baseline
- T2:Observational (Questionnaire): Patients with complete questionnaires to assess financial burden at 12 months
Arm/Group | T0: Observational (Questionnaire) | T2:Observational (Questionnaire)
Number analyzed (Participants) | 241 | 241
score on a scale | 23.5 (11.9) | 28.6 (11.7)
Statistical Analysis 1: Comparison: T0: Observational (Questionnaire) vs T2:Observational (Questionnaire); Age covariate effect on change in COST The linear (non-longitudinal) model of [change in COST from baseline to 12-month follow-up] included covariates for: age, Baseline COST score, cancer stage, cancer type, chemotherapy, comorbidities, education, FACT-G7, gender, income, marital status, insurance status, race, safety-net hospital, self-efficacy, NDI. Null: All estimates are equal; Test type: Equivalence — No margin of equivalence; p = 0.74, Regression, Linear — P value: For the categorical variable with more than 2 levels, this is the p value from the overall test of the null hypothesis that all estimates are equal against the alternative that at least one is different; Slope = 0, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 2: Comparison: T0: Observational (Questionnaire) vs T2:Observational (Questionnaire); Baseline COST effect on change in COST The linear (non-longitudinal) model of [change in COST from baseline to 12-month follow-up] included covariates for: age, Baseline COST score, cancer stage, cancer type, chemotherapy, comorbidities, education, FACT-G7, gender, income, marital status, insurance status, race, safety-net hospital, self-efficacy, NDI. Null: All estimates are equal; Test type: Equivalence — No margin of equivalence; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Slope = -0.4, 95% CI 2-sided [-0.6 to -0.3]
Statistical Analysis 3: Comparison: T0: Observational (Questionnaire) vs T2:Observational (Questionnaire); Cancer type (Colon cancer, Rectal cancer and Rectosigmoid) effect on change in COST The linear (non-longitudinal) model of [change in COST from baseline to 12-month follow-up] included covariates for: age, Baseline COST score, cancer stage, cancer type, chemotherapy, comorbidities, education, FACT-G7, gender, income, marital status, insurance status, race, safety-net hospital, self-efficacy, NDI. Null: All estimates are equal; Test type: Equivalence — No margin of equivalence; p = 0.002, Regression, Linear — This is the p value of the null hypothesis that COST estimates for all cancer types (Colon cancer, Rectal cancer and Rectosigmoid) are equal against the alternative that at least one is different
Statistical Analysis 4: Comparison: T0: Observational (Questionnaire) vs T2:Observational (Questionnaire); FACT-G7 effect on change in COST The linear (non-longitudinal) model of [change in COST from baseline to 12-month follow-up] included covariates for: age, Baseline COST score, cancer stage, cancer type, chemotherapy, comorbidities, education, FACT-G7, gender, income, marital status, insurance status, race, safety-net hospital, self-efficacy, NDI. Null: All estimates are equal; Test type: Equivalence — No margin of equivalence; p = 0.03, Regression, Linear; Slope = 0.3, 95% CI 2-sided [0.0 to 0.6]
Statistical Analysis 5: Comparison: T0: Observational (Questionnaire) vs T2:Observational (Questionnaire); Gender effect on change in COST The linear (non-longitudinal) model of [change in COST from baseline to 12-month follow-up] included covariates for: age, Baseline COST score, cancer stage, cancer type, chemotherapy, comorbidities, education, FACT-G7, gender, income, marital status, insurance status, race, safety-net hospital, self-efficacy, NDI. Null: All estimates are equal; Test type: Equivalence — No margin of equivalence; p = 0.13, Regression, Linear; Slope = 1.6, 95% CI 2-sided [-0.5 to 3.7]
Statistical Analysis 6: Comparison: T0: Observational (Questionnaire) vs T2:Observational (Questionnaire); RACE (White. Black Other) effect on change in COST The linear (non-longitudinal) model of [change in COST from baseline to 12-month follow-up] included covariates for: age, Baseline COST score, cancer stage, cancer type, chemotherapy, comorbidities, education, FACT-G7, gender, income, marital status, insurance status, race, safety-net hospital, self-efficacy, NDI. Null: All estimates are equal; Test type: Equivalence — No margin of equivalence; p = 0.91, Regression, Linear — This is the p value of the null hypothesis that COST estimates for all RACES (White, Black, other) are equal against the alternative that at least one is different
Statistical Analysis 7: Comparison: T0: Observational (Questionnaire) vs T2:Observational (Questionnaire); Neighborhood Deprivation (NDI) effect on change in COST The linear (non-longitudinal) model of [change in COST from baseline to 12-month follow-up] included covariates for: age, Baseline COST score, cancer stage, cancer type, chemotherapy, comorbidities, education, FACT-G7, gender, income, marital status, insurance status, race, safety-net hospital, self-efficacy, NDI. Higher NDI = greater neighborhood deprivation; Test type: Equivalence — No margin of equivalence; p > 0.99, Regression, Linear; Slope = 0.0, 95% CI 2-sided [-0.3 to 0.3]

2. Secondary Outcome: Reported Access and Utilization of Financial Services
Description: Will evaluate reported access and utilization of financial services (i.e. financial counselor, navigator, social workers) and its association to financial burden in the first 12 months after diagnosis of colon or rectal cancer treated with curative-intent. Will be assessed by Consumer Based Cancer Care Value Index (CCVI). For the continuous item variable, will conduct the paired t test to examine the difference if the distribution is normal. If not normally distributed, Wilcoxon signed rank test will be used. For the categorical item variable, the paired proportion test (e.g., McNemar test) will be used instead. The association between CCVI and COST measures will be evaluated using the Pearson or Spearman correlation coefficient.
Time Frame: Up to 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in Level of Self-reported Employment Limitations
Description: Change in level of self-reported employment limitations from baseline to 6, 12 and 24 months after study registration will be assessed by Work Productivity and Activity Impairment Questionnaire for a Specific Health Problem (WPAI:SHP). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows:
  Questions:
  1. = currently employed
  2. = hours missed due to specified problem
  3. = hours missed other reasons
  4. = hours actually worked
  5. = degree problem affected productivity while working
  6. = degree problem affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages.
  Percent work time missed due to problem: Q2/(Q2+Q4)
  Percent impairment while working due to problem: Q5/10
  Percent overall work impairment due to problem:
  Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)]
  Percent activity impairment due to problem: Q6/10
Time Frame: Baseline, 6, 12, and 24 months after cancer diagnosis
Measure: Mean (Standard Deviation); unit: percentage of activity impaired
Groups:
- Baseline Questionnaire: Patient questionnaires completed at baseline
- 6-month Questionnaire: Patient questionnaires completed at 6 months after cancer diagnosis.
- 12-month Questionnaire: Patient questionnaires completed at 12 months after cancer diagnosis.
- 24-month Questionnaire: Patient questionnaires completed at 24 months after cancer diagnosis.
Arm/Group | Baseline Questionnaire | 6-month Questionnaire | 12-month Questionnaire | 24-month Questionnaire
Number analyzed (Participants) | 192 | 69 | 60 | 57
percentage of activity impaired
  Work Time Missed | 39.7 (39.3) | 18.2 (30.7) | 4.8 (16.1) | 6.1 (18.0)
  Impairment of Activities at Work | 20.8 (33.4) | 28.1 (33.0) | 14.0 (24.6) | 14.4 (22.3)
  Overall Work Impairment | 51.8 (37.5) | 36.6 (36.6) | 17.8 (28.0) | 19.1 (26.8)
  Impairment of Activities Outside of Work | 33.2 (31.8) | 31.3 (31.9) | 17.0 (25.8) | 15.8 (24.2)
Statistical Analysis 1: Comparison: Baseline Questionnaire vs 6-month Questionnaire; Work Time Missed from Baseline to 6 Months; Test type: Equivalence — no margin; p = 0.4142, McNemar — alpha=0.05
Statistical Analysis 2: Comparison: Baseline Questionnaire vs 6-month Questionnaire; Impairment of Activities at Work from Baseline to 6 Months; Test type: Equivalence — no margin; p = 0.1797, McNemar
Statistical Analysis 3: Comparison: Baseline Questionnaire vs 6-month Questionnaire; Overall Work Impairment from Baseline to 6 Months; Test type: Equivalence — no margin; p = 0.8415, McNemar
Statistical Analysis 4: Comparison: Baseline Questionnaire vs 6-month Questionnaire; Impairment of Activities Outside of Work from Baseline to 6 Months; Test type: Equivalence — no margin; p = 0.6831, McNemar
Statistical Analysis 5: Comparison: Baseline Questionnaire vs 12-month Questionnaire; Work Time Missed from Baseline to 12 Months; Test type: Equivalence — no margin; p < .0001, McNemar
Statistical Analysis 6: Comparison: Baseline Questionnaire vs 12-month Questionnaire; Impairment of Activities at Work from Baseline to 12 Months; Test type: Equivalence — no margin; p = 0.0455, McNemar
Statistical Analysis 7: Comparison: Baseline Questionnaire vs 12-month Questionnaire; Overall Work Impairment from Baseline to 12 Months; Test type: Equivalence — no margin; p < .0001, McNemar
Statistical Analysis 8: Comparison: Baseline Questionnaire vs 12-month Questionnaire; 3 Impairment of Activities Outside of Work from Baseline to 12 Months; Test type: Equivalence — no margin; p = 0.0164, McNemar
Statistical Analysis 9: Comparison: Baseline Questionnaire vs 24-month Questionnaire; Work Time Missed from Baseline to 24 Months; Test type: Equivalence — nomargin; p = 0.0027, McNemar
Statistical Analysis 10: Comparison: Baseline Questionnaire vs 24-month Questionnaire; Impairment of Activities at Work from Baseline to 24 Months; Test type: Equivalence — no margin; p = 0.0124, McNemar
Statistical Analysis 11: Comparison: Baseline Questionnaire vs 24-month Questionnaire; Overall Work Impairment from Baseline to 24 Months; Test type: Equivalence — no margin; p < .0001, McNemar
Statistical Analysis 12: Comparison: Baseline Questionnaire vs 24-month Questionnaire; Impairment of Activities Outside of Work from Baseline to 24 Months; Test type: Equivalence — no margin; p = 0.0011, McNemar

4. Secondary Outcome: Level of Self-reported Employment Limitations (Dichotomized)
Description: Change in level of self-reported employment limitations from baseline to 6, 12 and 24 months after study registration will be assessed by Work Productivity and Activity Impairment Questionnaire for a Specific Health Problem (WPAI:SHP). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. These outcomes were further dichotomized at 50%, such that Impairment > 50% was considered impaired and Impairment <=50% was not-impaired
Time Frame: Baseline, 6, 12, and 24 months after cancer diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Questionnaire | 6-month Questionnaire | 12-month Questionnaire | 24-month Questionnaire
Number analyzed (Participants) | 192 | 69 | 60 | 57
Participants
  Work Time Missed: Impaired ( score >50%) | 124 | 55 | 58 | 54
  Work Time Missed: Impaired ( score <=50%) | 68 | 14 | 2 | 3
  Impairment of Activities at Work: Impaired ( score >50%) | 139 | 47 | 51 | 49
  Impairment of Activities at Work: Impaired ( score <=50%) | 53 | 22 | 9 | 8
  Overall Work Impairment: Impaired ( score >50%) | 93 | 40 | 49 | 47
  Overall Work Impairment: Impaired ( score <=50%) | 99 | 29 | 11 | 10
  Impairment of Activities Outside of Work: Impaired ( score >50%) | 121 | 47 | 49 | 48
  Impairment of Activities Outside of Work: Impaired ( score <=50%) | 71 | 22 | 11 | 9

5. Secondary Outcome: Long Term Outcomes After Diagnosis for Adherence
Description: Will evaluate long term outcomes at 24 months after diagnosis for adherence to clinical follow-up guidelines. Specially, linear (or generalized linear) mixed model will be fit to study the change in the mean response over time. In case the changes in the mean response over time are not linear, the quadratic trends or non-linear trends via spline may be considered in the modeling. Interactions will be evaluated as well.
Time Frame: At 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Long Term Outcomes After Diagnosis for Financial Burden
Description: Will evaluate long term outcomes at 24 months after diagnosis for financial burden. Specially, linear (or generalized linear) mixed model will be fit to study the change in the mean response over time and also the effects of cancer type, stage, treatment plan and demographics, etc. on financial burden. In case the changes in the mean response over time are not linear, the quadratic trends or non-linear trends via spline may be considered in the modeling. Interactions will be evaluated as well.
Time Frame: At 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Long Term Outcomes After Diagnosis for Employment Limitations
Description: Will evaluate long term outcomes at 24 months after diagnosis for employment limitations. Specially, linear (or generalized linear) mixed model will be fit to study the change in the mean response over time. In case the changes in the mean response over time are not linear, the quadratic trends or non-linear trends via spline may be considered in the modeling. Interactions will be evaluated as well.
Time Frame: At 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Change of Quality-of-life (QoL) Outcome
Description: Will evaluate the change of QoL from baseline to 12 months and its association with predictors. Will be evaluated by Functional Assessment of Cancer Therapy-General.
Time Frame: Baseline up to 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Changes Self-reported Financial Burden Between Baseline and 12 Month [EORTC]
Description: Financial Burden was evaluated using a single item from European Organization for Research and Treatment of Cancer Questionnaire 30 [EORT30]) with responses for both baseline and 12 months
  EORTC30 question:
  Has your physical condition or medical treatment caused you financial difficulties?
  * Not at all
  * A little
  * Quite a bit
  * Very much with higher values indicating greater financial difficulty (burden) Responses were dichotomized into No difficulty ("Not at All" ) and some difficulty ( "A little", "Quite a bit", or "Very much")
Time Frame: Baseline and12 months
Population: participants who completed both the baseline and 12 month EORTC questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- No Difficulty ("Not at All" ) at Baseline: This group represents the participants who responded "Not at All" to the EORTC30 question:
  Has your physical condition or medical treatment caused you financial difficulties?
  * Not at all
  * A little
  * Quite a bit
  * Very much
- Some Difficulty ( "A Little", "Quite a Bit", or "Very Much") at Baseline: This group represents the participants who responded "A little", "Quite a bit", or "Very much" to the EORTC 30 question:
  Has your physical condition or medical treatment caused you financial difficulties?
  * Not at all
  * A little
  * Quite a bit
  * Very much
Arm/Group | No Difficulty ("Not at All" ) at Baseline | Some Difficulty ( "A Little", "Quite a Bit", or "Very Much") at Baseline
Number analyzed (Participants) | 91 | 114
Participants
  No difficulty ("Not at All" ) at 12 months | 74 | 34
  Some Difficulty ( "A little", "Quite a bit", or "Very much") at 12 Months | 17 | 80
Statistical Analysis 1: Comparison: No Difficulty ("Not at All" ) at Baseline vs Some Difficulty ( "A Little", "Quite a Bit", or "Very Much") at Baseline; the McNemar test was used to compare the results assuming a null of no difference; Test type: Equivalence — no equivalence margin was assumed; p = 0.017, McNemar

ADVERSE EVENTS:
Time Frame: up to 24 months
Description: This is an observational study which only collected All-Cause Mortality and Serious Adverse Events, other adverse event data was not collected
Groups:
- Before Completing Any Questionaire: Patients registered for participation but off study before completing any study questionnaire:
  Quality-of-Life Assessment: Ancillary studies Questionnaire Administration: Ancillary studies
- Observational (Questionnaire) Baseline Questionnaire: All Patients complete questionnaires over 20-60 minutes after cancer diagnosis at baseline
  Quality-of-Life Assessment: Ancillary studies Questionnaire Administration: Ancillary studies
- Observational (Questionnaire) 3 Months: All Patients complete questionnaires over 20-60 minutes at 3 months after cancer diagnosis.
  Quality-of-Life Assessment: Ancillary studies Questionnaire Administration: Ancillary studies
- Observational (Questionnaire) 6 Months: All Patients complete questionnaires over 20-60 minutes at 6 months after cancer diagnosis.
  Quality-of-Life Assessment: Ancillary studies Questionnaire Administration: Ancillary studies
- Observational (Questionnaire) 12 Months: All Patients complete questionnaires over 20-60 minutes at 12 months after cancer diagnosis.
  Quality-of-Life Assessment: Ancillary studies Questionnaire Administration: Ancillary studies
- Observational (Questionnaire) 24 Months: All Patients complete questionnaires over 20-60 minutes at 24 months after cancer diagnosis.
  Quality-of-Life Assessment: Ancillary studies Questionnaire Administration: Ancillary studies
Arm/Group | Before Completing Any Questionaire | Observational (Questionnaire) Baseline Questionnaire | Observational (Questionnaire) 3 Months | Observational (Questionnaire) 6 Months | Observational (Questionnaire) 12 Months | Observational (Questionnaire) 24 Months
All-Cause Mortality (participants affected / at risk) | 13/57 | 0/455 | 5/301 | 5/272 | 4/233 | 2/245
Serious Adverse Events (participants affected / at risk) | 13/57 | 0/455 | 4/301 | 4/272 | 12/233 | 2/245
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Before Completing Any Questionaire (N=57) | Observational (Questionnaire) Baseline Questionnaire (N=455) | Observational (Questionnaire) 3 Months (N=301) | Observational (Questionnaire) 6 Months (N=272) | Observational (Questionnaire) 12 Months (N=233) | Observational (Questionnaire) 24 Months (N=245)
Death Nos (General disorders) | 13 (13) | 0 (0) | 4 (4) | 4 (4) | 12 (12) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03516942/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03516942/ICF_001.pdf